CLINICAL TRIAL: NCT05848102
Title: Dapagliflozin Effect on FunctiOnal Mitral Regurgitation and Myocardial Fibrosis (DEFORM): a Multicenter Randomized Controlled Trial
Brief Title: Dapagliflozin Effect on FunctiOnal Mitral Regurgitation and Myocardial Fibrosis (DEFORM)
Acronym: DEFORM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); Jieyang People's Hospital (Other); Eighth Affiliated Hospital, Sun Yat-sen University (Other); Affiliated Hospital of Guangdong Medical University (Other); Yuebei People's Hospital (Other); Zhongshan People's Hospital, Guangdong, China (Other)
Responsible Party: Principal Investigator, Xiao-dong Zhuang, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DEFORM Study
Record Dates: First submitted 2023-04-13; First posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-04

CONDITIONS: Functional Mitral Regurgitation
Keywords: dapagliflozin; Guideline directed medical therapy
MeSH Terms: interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin arm (Experimental): In the Dapagliflozin arm, participants with functional mitral regurgitation of more than moderate and left ventricular ejection fraction of more than 40% will add oral drug of Forxiga (Dapagliflozin, specification: 10mg) of 10 mg per day on the basis of regular guideline directed medical therapy for functional mitral regurgitation for 6 months.
  Interventions: Drug: dapagliflozin
- GDMT arm (No Intervention): In the guideline directed medical therapy (GDMT) arm, participants with functional mitral regurgitation of more than moderate and left ventricular ejection fraction of more than 40% will continue to maintain the original treatment of GDMT for 6 month.

INTERVENTIONS:
Drug: dapagliflozin — FORXIGA（Dapagliflozin Tablets), manufacturer/marketer: AstraZeneca, salt composition: Dapagliflozin (10mg), one tablet once and once a day.
  Arms: Dapagliflozin arm

SUMMARY:
The goal of this clinical trial is to learn about the effect of dapagliflozin on reducing the degree of mitral regurgitation and myocardial fibrosis in patients with functional mitral regurgitation (FMR) of more than moderate and left ventricular ejection fraction (LVEF) more than 40%.

The main question[s] it aims to answer are:

* For FMR patients with EF>40%, whether adding SGLT2 to guideline directed medical therapy (GDMT) can reduce MR degree and myocardial fibrosis, as well as improve patient's cardio-pulmonary function and quality of life is unknown.
* For FMR patients with EF>40%, whether adding SGLT2 to GDMT can decelerate the progression of FMR to end-stage heart failure, reduce the demand for percutaneous mitral valve repair and improve the prognosis is unknown.

Participants in dapagliflozin arm will add dapagliflozin of 10 mg/d orally for 6 months on the basis of regular GDMT for FMR. Researchers will compare the dapagliflozin arm to the GDMT arm who only accept the regular GDMT to see if the effective regurgitant orifice area was decreased.

The primary endpoint was the effective regurgitant orifice area(EROA) change from baseline to 6 months.

The secondary endpoints include the cardiac magnetic resonance assessment of myocardial fibrosis, the N-terminal fragment of the pro brain natriuretic peptides(NT-pro BNP), maximal exercise capacity by cardiopulmonary exercise testing, distance in the 6 minutes walking test, Kansas City cardiomyopathy questionnaire and Cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to get enrolled;
2. Age 18-90 years old, gender is not limited;
3. More than moderated FMR ( EROA by echocardiography ≥0.2cm2) , and LVEF more than 40%;
4. The structure of mitral valve leaflets and chordae is normal;
5. GDMT for FMR has been taken orally for more than 2 weeks, and the dose has not been adjusted for more than 2 weeks (If there is no contraindication, the drugs includes β blockers, the renin-angiotensin system inhibitors [Angiotensin-Converting Enzyme Inhibitors/Angiotensin Receptor Blockers/angiotensin receptor neprilysin inhibitor], aldosterone receptor antagonists), and for the last 2 weeks no intravenous drug for heart failure were used.

Exclusion Criteria:

1. Have indication for dapagliflozin;
2. Angioedema, or allergic to dapagliflozin;
3. Already taking Dapagliflozin or other SGLT2 inhibitors;
4. Primary mitral valve structural damage, such as rheumatic heart disease, mitral valve prolapse;
5. Non-dialysis patients with estimated glomerular filtration rate<30ml/min/1.73m2;
6. Dialysis patients;
7. Acute myocardial infarction, acute myocarditis, or percutaneous transluminal coronary intervention, coronary artery bypass grafting and other vascular reconstruction operations have occurred within 3 months;
8. Those who plan to take vascular reconstruction, cardiac resynchronization therapy, percutaneous mitral valve repair, surgical valve repair or replacement within 3 months after enrollment;
9. Complications of obvious aortic valve disease (more than moderate stenosis or more than moderate regurgitation);
10. Thyroid function combined with hyperthyroidism has not returned to normal;
11. Pregnant and lactating women.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2022-12-23 (Actual); Primary Completion 2024-10-23 (Estimated); Study Completion 2025-04-23 (Estimated)

PRIMARY OUTCOMES:
Mitral valve effective regurgitant orifice area change | From baseline to 6 month
  Evaluated by echocardiography at baseline and 6 month

SECONDARY OUTCOMES:
myocardial fibrosis change | from baseline to 6 month
  Evaluated by cardiac magnetic resonance
NT-proBNP change | from baseline to 6 month
  N-terminal pro-brain natriuretic peptide(NT-proBNP) tested in Venous blood sample
KCCQ-12 score | from baseline to 6 month
  Cardiomyopathy questionnaire (Kansas City):(KCCQ-12)
cardiopulmonary exercise testing score | from baseline to 6 month
  Cardiorespiratory functional assessment
Distance of 6 minutes walking test | from baseline to 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Zhuang, PhD, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (3):
- China (3):
  - The Third Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University, Guanzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No